CLINICAL TRIAL: NCT02497443
Title: Phase 1 Study of Autologous Mesenchymal Stem Cell Application for Therapy of Drug-Resistant Symptomatic Epilepsy
Brief Title: Safety of Autologous MSC Infusion to Treat Epilepsy
Acronym: AMSCDRSE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ministry of Public Health, Republic of Belarus (Other Government)
Responsible Party: Principal Investigator, Potapnev Michael, MD, Prof., Head the Department of Cellular BioTechnologies, Republican Scientific and Practical Center of Transfusiology and Medical Biotechnologies, Ministry of Public Health, Republic of Belarus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Minsk-MH001
Record Dates: First submitted 2015-04-07; First posted 2015-07-14 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy
Keywords: drug-resistant symptomatic epilepsy; seizure; autologous mesenchymal stem cells; safety; remission; electroencephalography; refractory symptomatic epilepsy; autologous MSC; efficacy
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Masking was specified as Opel Label study in old format
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Pts undergoing carbamazepine, valproic acid, topiramate, lamotrigine, or phenobarbital (i.e.anti-epileptic drugs [AEDs]) and receiving autologous mesenchymal stem cells
  Interventions: Biological: Autologous mesenchymal stem cells
- control group (No Intervention): Pts undergoing carbamazepine, valproic acid, topiramate, lamotrigine, or phenobarbital (i.e.AEDs)

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — Autologous bone marrow-derived mesenchymal stem cells, expanded ex vivo and neuroinduced (a portion of the cells). The final autologous cultured MSCs (0.7 -1.4 x 106 cells/kg of weigh) and autologous neuroinduced MSCs (0.04 - 0.1 x 106 cells/kg of weigh) were used for intravenous administration (cultured MSCs) and a subsequent endolumbal injection (neuroinduced MSCs) one week later in the patients in an autologous manner.
  Arms: study group

SUMMARY:
• The goal of this study was to evaluate the safety and efficacy of autologous MSC application for the therapy of drug-resistant symptomatic epilepsy. Adult (18-60 years old) patients (pts) of both sexes suffering from refractory epilepsy with frequent (>5 events per month) seizures were included in this study. The pts were randomized to the standard treatment with anti-epileptic drugs (control group, 30 pts) or anti-epileptic drugs plus autologous mesenchymal stem cells (MSCs) (study group, 30 pts). The pts in the study group received one intravenous injection of ex vivo expanded MSCs (40-101 x 106 cells) and one subsequent endolumbal injection of neuroinduced MSCs (2.7 - 8.0 x 106 cells). Both the unfavorable reactions to MSC infusions and the clinical effects, including complications, were examined. The unfavorable reactions to the MSC injections included local pain or hemorrhage at the site of injection and systemic reactions of the central nervous system (CNS; i.e., hyperthermia, fatigue, and myalgia).The possible beneficial effects of therapy in the two groups of pts were examined based on clinical observations and electroencephalography measurements (prior and 12 months after the application of the MSC-based therapy). To determine potential changes in disease progression, the signs of cognitive impairment, behavioral disorders, and particularly, changes in seizure character and frequency were evaluated using the National Hospital Scale of Seizure Severity. The main points of disease monitoring were "yes" or "no" responses (to therapy), seizure frequency (per month), and remission of disease. Electroencephalography (EEG) recordings were performed to evaluate electrical alpha, beta, theta and delta waves based on standard and additional criteria. The paroxismality index, the peak frequency of EEG activity, the index of slow activity, and the summarized points of EEG pathology signs were calculated for each patient. All assessments were performed for the pts in the control and study groups, and the obtained data were compared to identify the potential differences between the two pts groups. Therapy was terminated when immediate unfavorable reactions to the MSC injections were observed. The final observation of each patient included clinical and EEG assessments at the time point of 12 months (or more) after the application of the MSC-based therapy.

DETAILED DESCRIPTION:
The main goal of this phase 1 clinical trial was to evaluate the safety of an autologous mesenchymal stem cell (MSC) application as therapy for drug-resistant symptomatic epilepsy in a one-center study. It is well known that drug-resistant symptomatic epilepsy is a dramatically invalidating disorder for which applied stationary and outpatient therapies have no real clinical effect. Therefore new approaches are needed to reach remission, to stop disease progression, and to increase patient quality of life. For this study, adult (18-60 years old) patients (pts) of both sexes suffering from drug-resistant symptomatic epilepsy with frequent (>5 events per month) seizures were included into study. Drug-resistance was defined by a lack of any evident clinical response (i.e., no decrease in seizure frequency or reduction in disease progression) of the pts with symptomatic epilepsy to carbamazepine, valproic acid, topiramate, lamotrigine, or phenobarbital (i.e., anti-epileptic drugs[AEDs]) as monotherapies and in different combinations over the previous one calendar year. The criteria for exclusion were patient refusal to participate, unfavorable reactions to therapy, CNS inflammatory conditions, chronic psychoses, CNS tumors, relapses of chronic somatic or neurologic diseases, and blood positivity for hepatitis B or C or HIV. The plan included the inclusion of 30 pts in the study group and 30 pts in the control group over a period of 5 years. The pts were randomized to standard treatment with AEDs (control group) or AEDs plus autologous mesenchymal stem cells (MSCs, study group). The MSCs were obtained from bone marrow samples of the same patient and were purified and expanded ex vivo in a specialized cellular biotechnology laboratory. The MSCs were characterized by immunophenotyping as CD90+CD105 +CD45-CD34-cells. After 3 weeks of cultivation in vitro, a portion of the MSC were additionally cultured for 7 days in Neurocult-XF proliferation medium to obtain neuroinduced MSCs. Neuroinduction was proved by the presence of the genetic markers nestin and neuron-specific enolase. Finally, 40-101 x 106 autologous cultured MSCs and 2.7 - 8.0 x 106 autologous neuroinduced MSCs were harvested, resuspended in saline solution containing 5% autologous blood serum for injection, and, following a measurement of the viability (98% cells), transferred to the clinical center.

The pts in the study group received one slowly delivered (over 5-10 minutes) intravenous injection of ex vivo expanded autologous MSCs in a volume of 20 ml, and 5-7 days later, each patient in the study group received an additional slowly delivered endolumbal injection of the neuroinduced MSCs in a volume of 5 ml. Both unfavorable reactions to the MSC injections (over one day following the performance of the procedures) and the early (up to one month) and late (up to 6 months) clinical effects, including complications, were evaluated. Unfavorable reactions to the MSC injections included local pain or hemorrhage at the site of injection and systemic reactions of the central nervous system (CNS, i.e., hyperthermia, fatigue, and myalgia). Later potential unfavorable systemic reactions of the CNS and vascular system, including infectious and noninfectious complications of the progression of the disease to be controlled, were examined. All of the events were documented in medical cards. In cases in which these events exhibited dangerous characteristics, they were declared to members of the monitoring board (the center's ethical committee) for the evaluation of the exclusion of the patients from the study or the termination of the clinical study.

Also evaluated were the possible beneficial effects of MSC-based therapy in the pts of the study group. These effects were detected via clinical observations at selected therapy time points (i.e., 3 and 12 months after the application of the MSC-based therapy) and electroencephalography measurements prior to and one year after the therapy. To determine the possible changes in disease progression, signs of cognitive impairment, behavioral disorders, and changes in seizure characteristics and frequency were evaluated. For the evaluation of cognitive impairment, we used the Mini-Mental State Examination. The handicapping effect of disease on daily life was scoring using the Subjective Handicap of Epilepsy Scale. State anxiety and depression were evaluated using the Hospital anxiety and depression scale . Changes in seizure characteristics and frequency were evaluated using the National Hospital Scale of Seizure Severity. The processes of voluntary attention and performance were studied with Schulte tables according to the methods of Kraepelin. Schulte tables were used to study sensorimotor reaction times and the distribution and stability of attention. The "Account of Kraepelin" method was used to study health, fatigue and the stability of attention. The assessment of short-term memory was performed via the method of memorizing 10 words; this method aims to determine the volume and speed of oral-aural memory.

Main clinical characteristics that are used for disease monitoring were "yes" or "no" responses (regarding therapy), seizure frequency (per month), and remission of disease at the early (3 months) and late (12 month and more) time points after therapy. To evaluate partial responses to therapy, the numbers of pts who exhibited 50% reductions in seizure frequency were assessed. Seizure type (i.e., generalized tonic-clonic, partial complex, simple partial, and multiple types of seizures) was also evaluated along with changes in seizure type during the treatment course.

Electroencephalography recordings were performed at admission and across the monitoring period using a Mizar EEG 201 encephalography system with biopotential registration from 16 body points according to the "10-20" scheme. The observed electrical alpha, beta, theta and delta waves were analyzed in 3-min segments (with further recalculation for each 1-minute segment) prior to (at admission) and 1 year after MSC application. The peak frequency of the alpha waves was also calculated. Both the spontaneous state and the state after the loading probe (hyperventilation and photostimulation) were evaluated for each patient. The characteristics of the electroencephalographies (EEG) were attributed to local and diffuse cortical alterations. We evaluated the paroxysmality index, quantities of local and generalized spikes of epileptiform waves per minute, peak frequency of EEG activity, index of slow activity, and summarized points of EEG pathology signs. EEGs with epileptiform activity included spikes, spike-slow waves, and high-amplitude spikes. The EEG recordings were performed based on standard and additionally proposed criteria . All of the assessments were performed for the pts in the control and study groups, and the obtained data were compared to determine the potential differences due to the additionally performed MSC-based therapy. A patient's therapy was terminated at any time point if immediate unfavorable reactions to the MSC injections were observed. The final observations of the patients included clinical and EEG assessments at 12 months (or more) after the application of the MSC-based therapy. The summarized data for the pts in the control and study groups were collected in an electronic database for further analysis and interpretations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic epilepsy,
* Disease progression for the last 1-3 years,
* Resistance of epilepsy to therapy with carbamazepine, valproic acid, topiramate, lamotrigine, and phenobarbital (anti-epileptic drugs/AEDs) as monotherapies or combination therapies;
* Signed informed consent

Exclusion Criteria:

* Central nervous system inflammatory disorders (meningoencephalitis of viral or parasite origin),
* Chronic decompensated psychoses ,dementia, social disadaptation,
* Central nervous system tumours.
* Blood positivity for hepatitis B or C or HIV infection;
* According to the judgment of the researchers, subjects who were unable to complete the study or may not have been able to comply with the requirements of this study (due to administrative or other reasons).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Safety of autologous bone marrow-derived Mesenchymal Stem Cells in patients with Drug-Resistant Symptomatic Epilepsy | 360 days
  * vital signs
  * adverse events related to infusion
  * physical examination indexes

SECONDARY OUTCOMES:
Efficacy of autologous bone marrow-derived Mesenchymal Stem Cells in patients with Drug-Resistant Symptomatic Epilepsy | 360 days
  * Complete (remission), partial response (>50% reduction of seizure) rate at 90 and 360 days
  * Complete response(CR)rate (%)=(number of CR/number of participants)*100%
  * Partial response(PR)rate (%)=(number of PR/number of participants)*100%

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Dakukina, MD,PhD, Principal Investigator — Deputy Director for Research, Republican Scientific and Practical Center for Mental Health, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) include patient code, date of birth, sex, history of disease, efficacy of stationary treatment with AED, list of descripted medicines, description of clinical state include types and frequency of seizures, paroxysmal spike-wave electroencephalography activity . Treatment outcome will be estimated at timepoint 12 months, additional timepoints for some parameters may be estimated at 3 and|or 6 months. The main outcome parameters are frequency and type of seizures, anxiety, depression, paroxysmal spike-wave EEG activity, NHS seizure severity score. Patient response to MSC-based cell therapy was estimated at 50% and 100% threshold in seizure frequency reduction.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Final Record and accepted data base of participants wil become available after finalization of study and will be available for one year
Access Criteria: Access will be available for physicians and researches, specialized in biomedical studies
URL: https://yadi.sk/i/vZT66BGKk-iYIw

REFERENCES:
- [Background] O'Donoghue MF, Duncan JS, Sander JW. The subjective handicap of epilepsy. A new approach to measuring treatment outcome. Brain. 1998 Feb;121 ( Pt 2):317-43. doi: 10.1093/brain/121.2.317. PMID 9549509
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Shakhbazau AV, Goncharova NV, Kosmacheva SM, Kartel' NA, Potapnev MP. Plasticity of human mesenchymal stem cell phenotype and expression profile under neurogenic conditions. Bull Exp Biol Med. 2009 Apr;147(4):513-6. doi: 10.1007/s10517-009-0547-6. English, Russian. PMID 19704961
- [Derived] Hlebokazov F, Dakukina T, Potapnev M, Kosmacheva S, Moroz L, Misiuk N, Golubeva T, Slobina E, Krasko O, Shakhbazau A, Hlavinski I, Goncharova N. Clinical benefits of single vs repeated courses of mesenchymal stem cell therapy in epilepsy patients. Clin Neurol Neurosurg. 2021 Aug;207:106736. doi: 10.1016/j.clineuro.2021.106736. Epub 2021 Jun 8. PMID 34119901
- [Derived] Hlebokazov F, Dakukina T, Ihnatsenko S, Kosmacheva S, Potapnev M, Shakhbazau A, Goncharova N, Makhrov M, Korolevich P, Misyuk N, Dakukina V, Shamruk I, Slobina E, Marchuk S. Treatment of refractory epilepsy patients with autologous mesenchymal stem cells reduces seizure frequency: An open label study. Adv Med Sci. 2017 Sep;62(2):273-279. doi: 10.1016/j.advms.2016.12.004. Epub 2017 May 10. PMID 28500900